CLINICAL TRIAL: NCT01688973
Title: Parallel (Randomized) Phase II Evaluation of ARQ 197 and ARQ 197 in Combination With Erlotinib in Papillary Renal Cell Carcinoma
Brief Title: Tivantinib With or Without Erlotinib Hydrochloride in Treating Patients With Metastatic or Locally Advanced Kidney Cancer That Cannot Be Removed by Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-01641; NCI-2012-01641 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); S1107; SWOG-S1107; S1107 (Other: SWOG); S1107 (Other: CTEP); U10CA180888 (NIH); U10CA032102 (NIH)
Record Dates: First submitted 2012-09-14; First posted 2012-09-20 (Estimated); Results first posted 2019-01-03 (Actual); Last update posted 2019-01-03 (Actual); Status verified 2018-12

CONDITIONS: Recurrent Renal Cell Carcinoma; Stage III Renal Cell Cancer; Stage IV Renal Cell Cancer; Type 1 Papillary Renal Cell Carcinoma; Type 2 Papillary Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Erlotinib Hydrochloride; ARQ 197

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (tivantinib) (Experimental): Patients receive tivantinib PO BID on days 1-28.
  Interventions: Other: Laboratory Biomarker Analysis; Drug: Tivantinib
- Arm II (tivantinib and erlotinib hydrochloride) (Experimental): Patients receive tivantinib PO BID and erlotinib hydrochloride PO QD on days 1-28.
  Interventions: Drug: Erlotinib Hydrochloride; Other: Laboratory Biomarker Analysis; Drug: Tivantinib

INTERVENTIONS:
Drug: Erlotinib Hydrochloride — 150 mg (1 tablet) by mouth on days 1-28, once daily, until disease progression
  Arms: Arm II (tivantinib and erlotinib hydrochloride)
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Tivantinib — 360 mg (3 tablets) by mouth, Twice daily (720 mg total daily dose) on days 1-28, until disease progression

SUMMARY:
This randomized phase II trial studies how well tivantinib with or without erlotinib hydrochloride works in treating patients with metastatic or locally advanced kidney cancer that cannot be removed by surgery. Tivantinib and erlotinib hydrochloride may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the response rate (confirmed complete and partial response) of patients with locally advanced or metastatic papillary renal cell carcinoma treated with either ARQ 197 (tivantinib) or ARQ 197 combined with erlotinib (erlotinib hydrochloride).

SECONDARY OBJECTIVES:

I. To assess the progression free survival (PFS) of patients with locally advanced or metastatic papillary renal cell carcinoma treated with either ARQ 197 or ARQ 197 combined with erlotinib.

II. To assess the safety and tolerability of ARQ 197 therapy and ARQ 197 combined with erlotinib.

III. To descriptively assess the role of prior treatment on outcome.

TERTIARY OBJECTIVES:

I. To bank tissue specimens for future use and once funding is obtained to evaluate the expression of tissue correlative biomarkers such as hepatocyte growth factor receptor (c-MET) and epidermal growth factor receptor (EGFR), and to perform exploratory correlation with clinical outcomes.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive tivantinib orally (PO) twice daily (BID) on days 1-28.

ARM II: Patients receive tivantinib PO BID and erlotinib hydrochloride PO once daily (QD) on days 1-28.

In both arms, courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 1 year and then every 6 months for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed papillary histology renal cell carcinoma which is metastatic, or locally advanced and unresectable; mixed histologies will be allowed provided that they contain >= 50% of the papillary component
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension; x-rays, scans or physical examinations used for tumor measurement must have been completed within 28 days prior to registration; x-rays, scans or physical examinations for non-measurable disease must have been completed within 42 days prior to registration; all disease must be assessed and documented on the Baseline Tumor Assessment form
* Patients with metastatic disease who have a resectable primary tumor and are deemed a surgical candidate may have undergone resection; at least 28 days must have elapsed since surgery and patient must have recovered from any adverse effects of surgery
* Patients with a history of brain metastases who are asymptomatic and have not received steroid therapy in the 14 days prior to registration are eligible; anti-seizure medications are allowed provided they are non-enzyme inducing (e.g. topiramate, levetiracetam, gabapentin)
* Patients may have received up to one prior systemic therapy for advanced or metastatic renal cell carcinoma; patients must not have received a MET inhibitor or erlotinib as prior therapy; at least 21 days must have elapsed since completion of prior systemic therapy, 42 days for nitrosoureas or mitomycin C; patients must have recovered from all associated toxicities at the time of registration
* Patients may have received prior radiation therapy, but must have measurable disease outside the radiation port; at least 21 days must have elapsed since completion of prior radiation therapy; patients must have recovered from all associated toxicities at the time of registration
* Patients must not be receiving or planning to receive any other investigational agents
* Patients must have a complete physical examination and medical history within 28 days prior to registration
* Patients must have a Zubrod performance status of 0-2
* White blood cell (WBC) >= 2,000/mcL
* Absolute neutrophil count (ANC) >= 1,000/mcL
* Platelet count >= 75,000/mcL
* Serum bilirubin =< 1.5 x institutional upper limits of normal (ULN)
* Serum glutamic oxaloacetic transaminase (SGOT)/aspartate aminotransferase (AST) and serum glutamic pyruvate transaminase (SGPT)/alanine aminotransferase (ALT) must be =< 1.5 x the institutional ULN unless the liver is involved with the tumor, in which case serum transaminase (SGOT/SGPT) must be =< 5 x the institutional ULN
* Serum creatinine must be =< 2 x the institutional ULN
* Sodium, potassium and calcium must be obtained within 14 days prior to registration
* Patients with a known history of the following corneal diseases are not eligible: dry eye syndrome, Sjogren's syndrome, keratoconjunctivitis sicca, exposure keratopathy, Fuchs' dystrophy or other active disorders of cornea
* Patients known to be human immunodeficiency virus (HIV)-positive and receiving combination anti-retroviral therapy are not eligible
* Patients must be able to take oral medications; patients must not have gastrointestinal tract disease resulting in an inability to take oral medication or a requirement for intravenous (IV) alimentation, prior surgical procedures affecting absorption, or active peptic ulcer disease; patients with intractable nausea or vomiting are not eligible
* Patients must not be pregnant or nursing; women/men of reproductive potential must have agreed to use an effective contraceptive method; a woman is considered to be of "reproductive potential" if she has had menses at any time in the preceding 12 consecutive months; in addition to routine contraceptive methods, "effective contraception" also includes heterosexual celibacy and surgery intended to prevent pregnancy (or with a side-effect of pregnancy prevention) defined as a hysterectomy, bilateral oophorectomy or bilateral tubal ligation; however, if at any point a previously celibate patient chooses to become heterosexually active during the time period for use of contraceptive measures outlined in the protocol, he/she is responsible for beginning contraceptive measures
* No other prior malignancy is allowed except for the following: adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, adequately treated stage I or II cancer from which the patient is currently in complete remission, or any other cancer from which the patient has been disease-free for 5 years
* Patients must be offered the opportunity to participate in specimen banking for future translational medicine studies
* All patients must be informed of the investigational nature of this study and must sign and give written informed consent
* As a part of the Oncology Patient Enrollment Network (OPEN) registration process the treating institution's identity is provided in order to ensure that the current (within 365 days) date of institutional review board approval for this study has been entered in the system

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2012-08-20; Primary Completion 2017-04-30 (Actual); Study Completion 2017-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Przemyslaw Twardowski, Principal Investigator — SWOG Cancer Research Network
Locations (214):
- United States (214):
  - University of Arizona Cancer Center-Orange Grove Campus, Tucson, Arizona
  - University of Arizona Cancer Center-North Campus, Tucson, Arizona
  - The University of Arizona Medical Center-University Campus, Tucson, Arizona
  - Kaiser Permanente-Anaheim, Anaheim, California
  - Kaiser Permanente-Baldwin Park, Baldwin Park, California
  - Kaiser Permanente-Bellflower, Bellflower, California
  - Alta Bates Summit Medical Center-Herrick Campus, Berkeley, California
  - Mills-Peninsula Medical Center, Burlingame, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Kaiser Permanente Hospital, Fontana, California
  - Kaiser Permanente - Harbor City, Harbor City, California
  - Kaiser Permanente-Irvine, Irvine, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Los Angeles County-USC Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - Kaiser Permanente-Cadillac, Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Fremont - Rideout Cancer Center, Marysville, California
  - Sutter Cancer Research Consortium, Novato, California
  - Stanford Cancer Institute, Palo Alto, California
  - Kaiser Permanente - Panorama City, Panorama City, California
  - Kaiser Permanente-Riverside, Riverside, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Kaiser Permanente-San Diego Mission, San Diego, California
  - Kaiser Permanente-San Diego Zion, San Diego, California
  - California Pacific Medical Center-Pacific Campus, San Francisco, California
  - Kaiser Permanente-San Marcos, San Marcos, California
  - Sutter Pacific Medical Foundation, Santa Rosa, California
  - Gene Upshaw Memorial Tahoe Forest Cancer Center, Truckee, California
  - Sutter Solano Medical Center/Cancer Center, Vallejo, California
  - Kaiser Permanente, Woodland Hills, California
  - University of Colorado Cancer Center - Anschutz Cancer Pavilion, Aurora, Colorado
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - George Washington University Medical Center, Washington D.C., District of Columbia
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Idaho Urologic Institute-Meridian, Meridian, Idaho
  - Hematology and Oncology Associates, Chicago, Illinois
  - Northwestern University, Chicago, Illinois
  - Hematology Oncology Associates of Illinois-Highland Park, Highland Park, Illinois
  - Hines Veterans Administration Hospital, Hines, Illinois
  - Presence Saint Mary's Hospital, Kankakee, Illinois
  - NorthShore Hematology Oncology-Libertyville, Libertyville, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Illinois Cancer Specialists-Niles, Niles, Illinois
  - Hematology Oncology Associates of Illinois - Skokie, Skokie, Illinois
  - Franciscan Saint Francis Health-Beech Grove, Beech Grove, Indiana
  - Franciscan Health Indianapolis, Indianapolis, Indiana
  - Reid Health, Richmond, Indiana
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Siouxland Regional Cancer Center, Sioux City, Iowa
  - Mercy Medical Center-Sioux City, Sioux City, Iowa
  - Saint Luke's Regional Medical Center, Sioux City, Iowa
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Saint Rose Ambulatory and Surgery Center, Great Bend, Kansas
  - Hays Medical Center, Hays, Kansas
  - Hutchinson Regional Medical Center, Hutchinson, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Providence Medical Center, Kansas City, Kansas
  - University of Kansas Cancer Center, Kansas City, Kansas
  - Cancer Center of Kansas-Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Cancer Center of Kansas-Liberal, Liberal, Kansas
  - Cancer Center of Kansas - McPherson, McPherson, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - Menorah Medical Center, Overland Park, Kansas
  - Saint Luke's South Hospital, Overland Park, Kansas
  - Cancer Center of Kansas - Parsons, Parsons, Kansas
  - Via Christi Hospital-Pittsburg, Pittsburg, Kansas
  - Kansas City NCI Community Oncology Research Program, Prairie Village, Kansas
  - Cancer Center of Kansas - Pratt, Pratt, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Salina Regional Health Center, Salina, Kansas
  - Saint Francis Hospital and Medical Center - Topeka, Topeka, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - Associates In Womens Health, Wichita, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas - Wichita, Wichita, Kansas
  - Via Christi Regional Medical Center, Wichita, Kansas
  - Wichita NCI Community Oncology Research Program, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - Michigan Cancer Research Consortium NCORP, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Beaumont Hospital-Dearborn, Dearborn, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Saint John Hospital and Medical Center, Detroit, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Genesys Regional Medical Center-West Flint Campus, Flint, Michigan
  - Genesys Regional Medical Center, Grand Blanc, Michigan
  - Allegiance Health, Jackson, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Sparrow Hospital, Lansing, Michigan
  - Saint Mary Mercy Hospital, Livonia, Michigan
  - Saint Joseph Mercy Oakland, Pontiac, Michigan
  - Lake Huron Medical Center, Port Huron, Michigan
  - Saint Mary's of Michigan, Saginaw, Michigan
  - Saint John Macomb-Oakland Hospital, Warren, Michigan
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Fairview-Southdale Hospital, Edina, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Metro Minnesota Community Oncology Research Consortium, Saint Louis Park, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Truman Medical Center, Kansas City, Missouri
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - North Kansas City Hospital, Kansas City, Missouri
  - Heartland Hematology and Oncology Associates Incorporated, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri
  - Saint Luke's East - Lee's Summit, Lee's Summit, Missouri
  - Liberty Radiation Oncology Center, Liberty, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Saint Joseph Oncology Inc, Saint Joseph, Missouri
  - Saint Louis Cancer and Breast Institute-South City, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Saint Louis-Cape Girardeau CCOP, St Louis, Missouri
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Nevada Cancer Research Foundation CCOP, Las Vegas, Nevada
  - Veterans Adminstration New Jersey Health Care System, East Orange, New Jersey
  - Glens Falls Hospital, Glens Falls, New York
  - Orange Regional Medical Center, Middletown, New York
  - Columbia University/Herbert Irving Cancer Center, New York, New York
  - University of Rochester, Rochester, New York
  - Kinston Medical Specialists PA, Kinston, North Carolina
  - Iredell Memorial Hospital, Statesville, North Carolina
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Columbus NCI Community Oncology Research Program, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - The Mark H Zangmeister Center, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital - Dayton, Dayton, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Samaritan North Health Center, Dayton, Ohio
  - Dayton NCI Community Oncology Research Program, Dayton, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Blanchard Valley Hospital, Findlay, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Saint Rita's Medical Center, Lima, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Southern Ohio Medical Center, Portsmouth, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - Greene Memorial Hospital, Xenia, Ohio
  - Genesis Healthcare System Cancer Care Center, Zanesville, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Geisinger Medical Center, Danville, Pennsylvania
  - Geisinger Medical Center-Cancer Center Hazleton, Hazleton, Pennsylvania
  - University of Pennsylvania/Abramson Cancer Center, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Geisinger Medical Group, State College, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Baylor University Medical Center, Dallas, Texas
  - Audie L Murphy Veterans Affairs Hospital, San Antonio, Texas
  - Cancer Therapy and Research Center at The UT Health Science Center at San Antonio, San Antonio, Texas
  - University Hospital, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - Cancer Care Center at Island Hospital, Anacortes, Washington
  - PeaceHealth Saint Joseph Medical Center, Bellingham, Washington
  - Harrison HealthPartners Hematology and Oncology-Bremerton, Bremerton, Washington
  - Highline Medical Center-Main Campus, Burien, Washington
  - Swedish Medical Center-Edmonds, Edmonds, Washington
  - Swedish Cancer Institute-Issaquah, Issaquah, Washington
  - Kadlec Clinic Hematology and Oncology, Kennewick, Washington
  - Skagit Valley Hospital, Mount Vernon, Washington
  - Harrison HealthPartners Hematology and Oncology-Poulsbo, Poulsbo, Washington
  - Harborview Medical Center, Seattle, Washington
  - Minor and James Medical PLLC, Seattle, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Group Health Cooperative-Seattle, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington
  - United General Hospital, Sedro-Woolley, Washington
  - Cancer Care Northwest - Spokane South, Spokane, Washington
  - Evergreen Hematology and Oncology PS, Spokane, Washington
  - Wenatchee Valley Hospital and Clinics, Wenatchee, Washington
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm I (Tivantinib): Patients receive tivantinib PO BID on days 1-28.
  Laboratory Biomarker Analysis: Correlative studies
  Tivantinib: Given PO
- Arm II (Tivantinib and Erlotinib Hydrochloride): Patients receive tivantinib PO BID and erlotinib hydrochloride PO QD on days 1-28.
  Erlotinib Hydrochloride: Given PO
  Laboratory Biomarker Analysis: Correlative studies
  Tivantinib: Given PO
Period: Overall Study
Arm/Group | Arm I (Tivantinib) | Arm II (Tivantinib and Erlotinib Hydrochloride)
Started | 27 | 28
Eligible/Evaluable Patients | 25 | 25
Completed | 25 | 25
Not Completed | 2 | 3
Not completed — Ineligible | 2 | 3

BASELINE CHARACTERISTICS:
Population: Two patients in Arm I and 3 patients in Arm II were ineligible and excluded from the analyses.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Tivantinib) | Arm II (Tivantinib and Erlotinib Hydrochloride) | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Continuous [Median (Full Range); unit: years] | 62.1 [20.3 to 76.1] | 63.6 [22.8 to 81.9] | 63.6 [20.3 to 81.9]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 10 | 16
  Male | 19 | 15 | 34
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 19 | 19 | 38
  Race: Black | 6 | 5 | 11
  Race: Unknown | 0 | 1 | 1
Histologic Grade [Count of Participants; unit: Participants] — The Fuhrman system ranges from 1-4; the higher the number, the more abnormal the cells look. A grade 1 cancer is usually slow growing. It is less likely to spread than a higher grade, such as a grade 4 cancer.
  Participants
    Unknown | 11 | 11 | 22
    1 | 0 | 0 | 0
    2 | 3 | 5 | 8
    3 | 7 | 6 | 13
    4 | 4 | 3 | 7
Histologic Subset [Count of Participants; unit: Participants]
  Pure Papillary | 20 | 23 | 43
  Mixed Histology | 5 | 2 | 7
Histologic Type [Count of Participants; unit: Participants] — Type 1 - lined by small cells with clear to basophilic cytoplasm; single layer of small oval nuclei; inconspicuous nucleoli; usually low grade (1 or 2) and low stage
  Type 2 - lined by large cells with abundant eosinophilic cytoplasm; large spherical nuclei; nuclei frequently pseudostratified or apical; usually high grade (3), many higher stage
  Participants
    Not Assigned | 12 | 14 | 26
    Type I | 2 | 1 | 3
    Type II | 11 | 10 | 21
Prior Nephrectomy [Count of Participants; unit: Participants]
  No | 4 | 7 | 11
  Yes | 21 | 18 | 39
Prior Systemic Therapy [Count of Participants; unit: Participants]
  None | 16 | 17 | 33
  One | 9 | 8 | 17
Performance Status [Count of Participants; unit: Participants] — Zubrod Performance Status Scale:
  0=Fully active, able to carry on all pre-disease performance without restriction.
  1. Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light housework, office work.
  2. Ambulatory and capable of self-care but unable to carry out any work activities; up and about more than 50% of waking hours.
  3. Capable of limited self-care, confined to bed or chair more than 50% of waking hours.
  4. Completely disabled; cannot carry on any self-care; totally confined to bed or chair.
  Participants
    0 | 12 | 9 | 21
    1 | 11 | 13 | 24
    2 | 2 | 3 | 5
    3 | 0 | 0 | 0
    4 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Response Rate (Confirmed Complete Response or Partial Response), Determined According to Response Evaluation Criteria in Solid Tumors
Description: Best Response is calculated from the sequence of objective statuses. CR: Two or more objective statuses of CR a minimum of four weeks apart documented before progression or symptomatic deterioration.
  PR: Two or more objective statuses of PR or better a minimum of four weeks apart documented before progression or symptomatic deterioration, but not qualifying as CR.
  Stable/no response: At least one objective status of stable/no response documented at least 6 weeks after registration and before progression or symptomatic deterioration, but not qualifying as anything else above.
  Increasing disease: Objective status of progression within 12 weeks of registration, not qualifying as anything else above.
  Symptomatic deterioration: Objective status of symptomatic deterioration within 12 weeks of registration, not qualifying as anything else above.
Time Frame: Up to 3 years
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Tivantinib) | Arm II (Tivantinib and Erlotinib Hydrochloride)
Number analyzed (Participants) | 25 | 25
Participants
  Complete Response | 0 | 0
  Partial Response | 0 | 0
  Stable/no response | 11 | 13
  Increasing disease | 14 | 7
  Symptomatic deterioration | 0 | 1
  Not Assessable | 0 | 4

2. Secondary Outcome: Frequency and Severity of Toxicities, Graded by the National Cancer Institute Common Terminology Criteria for Adverse Events Version 4.0
Description: This study utilized the CTCAE (NCI Common Terminology Criteria for Adverse Events) Version 4.0 for toxicity and Serious Adverse Event reporting. Patients were evaluated every two weeks for the first eight weeks and then once every four weeks. If all protocol treatment is delayed more than three weeks, patients were removed from protocol treatment
Time Frame: Up to 3 years
Population: All eligible patients who reported adverse events
Measure: Number; unit: Participants
Arm/Group | Arm I (Tivantinib) | Arm II (Tivantinib and Erlotinib Hydrochloride)
Number analyzed (Participants) | 25 | 25
Participants
  Alanine aminotransferase increased | 0 | 1
  Anemia | 2 | 1
  Aspartate aminotransferase increased | 0 | 1
  Dyspnea | 1 | 1
  Erythema multiforme | 0 | 1
  Fatigue | 0 | 1
  Febrile neutropenia | 0 | 1
  Hypertension | 1 | 0
  Hypoxia | 0 | 1
  Infections and infestations - Other, specify | 0 | 1
  Lung infection | 0 | 1
  Lymphocyte count decreased | 1 | 0
  Myocardial infarction | 0 | 1
  Nausea | 1 | 0
  Neutrophil count decreased | 1 | 0
  Pain in extremity | 1 | 0
  Pneumonitis | 0 | 1
  Rash acneiform | 0 | 2
  Rash maculo-papular | 0 | 1
  Stroke | 1 | 0
  Weight loss | 1 | 0
  White blood cell decreased | 1 | 1

3. Secondary Outcome: Progression-free Survival (PFS)
Description: From date of registration to date of first documentation of progression or symptomatic deterioration, or death due to any cause. Patients last known to be alive without report of progression are censored at date of last contact.
Time Frame: 30 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I (Tivantinib) | Arm II (Tivantinib and Erlotinib Hydrochloride)
Number analyzed (Participants) | 25 | 25
months | 2.0 [1.8 to 3.0] | 3.9 [1.8 to 7.3]

4. Other Pre Specified Outcome: Number of Participants With c-MET Amplification, Deletion and No Alteration
Time Frame: Baseline
Population: Tissue was only obtained from 35 patients. Exome of 16 patients were successfully sequenced using Agilent SureSelect probes.
  Arms were pooled due to no difference in response rate between the two arms
Measure: Count of Participants; unit: Participants
Groups:
- Pooled Arms: Pooled treatment arms for translational medicine objectives. Arms were pooled due to no difference in response rate between the two arms.
Arm/Group | Pooled Arms
Number analyzed (Participants) | 16
Participants
  Amplification | 6
  Deletion | 0
  No Alteration | 10

5. Other Pre Specified Outcome: Number of Participants With EGFR Amplification, Deletion and No Alteration
Time Frame: Baseline
Population: Tissue was only obtained from 35 patients. Exome of 16 patients were successfully sequenced using Agilent SureSelect probes.
Measure: Count of Participants; unit: Participants
Arm/Group | Pooled Arms
Number analyzed (Participants) | 16
Participants
  Amplification | 3
  Deletion | 1
  No Alteration | 12

ADVERSE EVENTS:
Time Frame: Up to 3 years
Description: This study utilized the CTCAE (NCI Common Terminology Criteria for Adverse Events) Version 4.0 for toxicity and Serious Adverse Event reporting. Patients were evaluated every two weeks for the first eight weeks and then once every four weeks. If all protocol treatment is delayed more than three weeks, patients were removed from protocol treatment.
  Adverse events and all-cause mortality is reported for all eligible patients.
Arm/Group | Arm I (Tivantinib) | Arm II (Tivantinib and Erlotinib Hydrochloride)
All-Cause Mortality (participants affected / at risk) | 20/25 | 21/25
Serious Adverse Events (participants affected / at risk) | 9/25 | 16/25
Other Adverse Events (participants affected / at risk) | 22/25 | 23/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Tivantinib) (N=25) | Arm II (Tivantinib and Erlotinib Hydrochloride) (N=25)
Anemia (Blood and lymphatic system disorders) | 1 | 2
Blood and lymphatic system disorders - Other (Blood and lymphatic system disorders) | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1
Atrial flutter (Cardiac disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 1 | 0
Cardiac disorders-Other (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1
Sinus bradycardia (Cardiac disorders) | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 2
Constipation (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 2
Fatigue (General disorders) | 1 | 2
Device related infection (Infections and infestations) | 0 | 1
Lung infection (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 2
Alkaline phosphatase increased (Investigations) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1
Blood bilirubin increased (Investigations) | 1 | 0
Platelet count decreased (Investigations) | 0 | 1
Weight loss (Investigations) | 1 | 0
White blood cell decreased (Investigations) | 0 | 1
Acidosis (Metabolism and nutrition disorders) | 0 | 2
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatremia (Metabolism and nutrition disorders) | 0 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Neoplasms benign, malignant and unspecified - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Dizziness (Nervous system disorders) | 0 | 1
Intracranial hemorrhage (Nervous system disorders) | 0 | 1
Stroke (Nervous system disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1
Hematuria (Renal and urinary disorders) | 1 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 | 1
Thromboembolic event (Vascular disorders) | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Tivantinib) (N=25) | Arm II (Tivantinib and Erlotinib Hydrochloride) (N=25)
Anemia (Blood and lymphatic system disorders) | 10 | 7
Sinus bradycardia (Cardiac disorders) | 2 | 4
Abdominal pain (Gastrointestinal disorders) | 4 | 4
Bloating (Gastrointestinal disorders) | 3 | 0
Constipation (Gastrointestinal disorders) | 5 | 4
Diarrhea (Gastrointestinal disorders) | 4 | 9
Flatulence (Gastrointestinal disorders) | 1 | 3
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2 | 1
Gastrointestinal disorders-Other (Gastrointestinal disorders) | 2 | 0
Mucositis oral (Gastrointestinal disorders) | 1 | 2
Nausea (Gastrointestinal disorders) | 11 | 14
Vomiting (Gastrointestinal disorders) | 3 | 6
Chills (General disorders) | 2 | 0
Edema limbs (General disorders) | 5 | 1
Fatigue (General disorders) | 13 | 13
Fever (General disorders) | 4 | 4
Flu like symptoms (General disorders) | 0 | 2
Localized edema (General disorders) | 1 | 2
Non-cardiac chest pain (General disorders) | 2 | 1
Pain (General disorders) | 4 | 2
Upper respiratory infection (Infections and infestations) | 2 | 1
Alanine aminotransferase increased (Investigations) | 2 | 5
Alkaline phosphatase increased (Investigations) | 3 | 4
Aspartate aminotransferase increased (Investigations) | 3 | 5
Blood bilirubin increased (Investigations) | 0 | 3
Creatinine increased (Investigations) | 6 | 6
Lymphocyte count decreased (Investigations) | 4 | 8
Neutrophil count decreased (Investigations) | 2 | 0
Weight gain (Investigations) | 3 | 2
Weight loss (Investigations) | 2 | 5
White blood cell decreased (Investigations) | 3 | 2
Anorexia (Metabolism and nutrition disorders) | 4 | 8
Hyperglycemia (Metabolism and nutrition disorders) | 7 | 8
Hyperkalemia (Metabolism and nutrition disorders) | 2 | 3
Hypoalbuminemia (Metabolism and nutrition disorders) | 4 | 4
Hypocalcemia (Metabolism and nutrition disorders) | 1 | 3
Hypokalemia (Metabolism and nutrition disorders) | 2 | 2
Hyponatremia (Metabolism and nutrition disorders) | 3 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 1
Chest wall pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 | 1
Dizziness (Nervous system disorders) | 2 | 1
Dysgeusia (Nervous system disorders) | 2 | 4
Headache (Nervous system disorders) | 2 | 2
Peripheral sensory neuropathy (Nervous system disorders) | 3 | 1
Anxiety (Psychiatric disorders) | 2 | 0
Depression (Psychiatric disorders) | 2 | 1
Insomnia (Psychiatric disorders) | 3 | 0
Hematuria (Renal and urinary disorders) | 0 | 2
Proteinuria (Renal and urinary disorders) | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 5
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 | 5
Alopecia (Skin and subcutaneous tissue disorders) | 5 | 2
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 3
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 2
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 | 13
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 | 3
Hypertension (Vascular disorders) | 4 | 6
Hypotension (Vascular disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-05-10): https://cdn.clinicaltrials.gov/large-docs/73/NCT01688973/Prot_SAP_000.pdf